CLINICAL TRIAL: NCT00795925
Title: Dose-Escalating Study of Propiverine Hydrochloride (Mictonetten®) in Children Suffering From Frequency-Urgency-Syndrome and Urinary Incontinence Indicative of Detrusor Overactivity (Overactive Bladder)
Brief Title: Dose-Escalating Study of Propiverine Hydrochloride in Children Suffering From Overactive Bladder
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: APOGEPHA Arzneimittel GmbH (Industry)
Masking: None
Other Study IDs: APOGEPHA-8403030
Record Dates: First submitted 2008-11-13; First posted 2008-11-21 (Estimated); Last update posted 2008-11-21 (Estimated); Status verified 2008-11

CONDITIONS: Overactive Bladder
Keywords: propiverine; anticholinergics; urinary incontinence; overactive bladder; children; dose-finding in children aged 5-10 years
MeSH Terms: conditions — Urinary Bladder, Overactive; Urinary Incontinence | interventions — propiverine

ARMS (1):
- propiverine hydrochloride (Experimental)
  Interventions: Drug: propiverine hydrochloride

INTERVENTIONS:
Drug: propiverine hydrochloride — coated tablets containing 5 mg
  consecutive dose escalation of 5 mg, 10 mg or 15 mg propiverine b.i.d.

SUMMARY:
The open-label dose-escalating two-centre study was designed to assess the pharmacokinetics as well as safety, tolerability and efficacy parameters of propiverine in patients 5-10 years of age suffering from frequency-urgency-syndrome and urinary incontinence indicative of detrusor overactivity (overactive bladder) for determination of the recommended dose in children.

ELIGIBILITY:
Main Inclusion Criteria:

* Micturition Frequency ≥6 micturitions during awake period
* Urge Incontinence Episodes ≥1/week
* Urgency Episodes ≥1/day

Main Exclusion Criteria:

* Contraindication to anticholinergic therapy
* Repeated measurement of Post Void Residual ≥20 mL
* Nocturnal Enuresis
* Clinically significant cardiovascular, hepatic, renal, gastrointestinal or hematological disease, psychiatric disorder or diabetes insipidus
* Anatomical abnormalities of the urinary tract

Ages: 5 Years to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 30 (Actual)
Dates: Start 2004-10; Study Completion 2005-12 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetic parameters of propiverine and its main metabolite propiverine N-oxide at steady state: Ctrough, Cmax, Tmax, AUC0-8h. Children were separated into 3 groups.

SECONDARY OUTCOMES:
Tolerability of propiverine. Efficacy: Changes from baseline: voiding frequency, incontinence and urgency episodes,voided volume. Safety: Post Void Residual (PVR),adverse events,laboratory values (urine, blood), ECG. | two weeks

CONTACTS AND LOCATIONS:
Overall Officials: Professor Ulla Sillen, M.D., Principal Investigator — Drottning Silvias ,Barn- och ungdomssjukhus, SU/Östra,416 85 Göteborg

REFERENCES:
- [Derived] Siegmund W, Sillen U, Lackgren G, Schnabel F, Murtz G, Feustel C. Pharmacokinetics and pharmacodynamics of propiverine in children aged between 5 and 10 years with symptoms of overactive bladder. Clin Pharmacokinet. 2010 May;49(5):335-42. doi: 10.2165/11319990-000000000-00000. PMID 20384395